CLINICAL TRIAL: NCT00733057
Title: A Double Blind Randomized Study of Minocycline for the Treatment of Negative and Cognitive Symptoms in Early-Phase Schizophrenia
Brief Title: Minocycline for the Treatment of Early-Phase Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Abarbanel Mental Health Center (Other Government)
Responsible Party: Dr. Yechiel Levkovitz, M.D., Shalvata Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMRI-GRANT-02T-244
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Negative and Cognitive Symptoms in Schizophrenia
Keywords: Minocycline; Schizophrenia; Negative symptoms; Cognitive
MeSH Terms: conditions — cyclopia sequence; Schizophrenia | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Minocycline treatment
  Interventions: Drug: Minocycline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (200 mg/day)

INTERVENTIONS:
Drug: Minocycline — Minocycline as an add-on drug (200 mg/day)
  Arms: 1
Drug: Placebo (200 mg/day)
  Arms: 2

SUMMARY:
Current antipsychotics have only a limited effect on two core symptoms of schizophrenia, negative symptoms and cognitive deficits. Minocycline is a second-generation tetracycline which has a beneficial effect in various neurological disorders. Recent findings in animal models and human case-reports suggest its potential for the treatment of these symptoms of schizophrenia. The current study aims to examine the efficacy of minocycline as add-on treatment for alleviating negative and cognitive symptoms in early-phase schizophrenia. The study will utilize a longitudinal double blind, randomized, placebo-controlled design with patients followed for six-months. Early-phase schizophrenia patients were recruited and randomly allocated to a minocycline or placebo treatment (2:1 ratio; 200 mg/day). The primary outcome measures are the Scale for Assessment of Negative Symptoms (SANS) and assessments of executive functions.

DETAILED DESCRIPTION:
Schizophrenia is a disorder characterized by disturbances in perception, thought, volition, socialization, psychomotor behavior and the sense of self. Although patients suffer from schizophrenia start from a point of relative normalcy or subtle impairment, following formal onset most patients experience, to some degree, clinical deterioration. This deterioration is manifest by the development of and increasing severity and persistence of psychotic and negative symptoms, cognitive impairment, and diminished social and functional capacity. The underlying causes of this clinical deterioration are not known, but is generally attributed to progression of the illness and associated with periods of active positive symptoms. The deterioration occurs primarily in the early stages of the illness and it is generally confined to the first 5 years after onset. It also does not progress in a linear fashion. Rather, after a period, patients stabilize at a level where they have persistent symptoms and are impaired in their social and vocational function. Despite the heterogeneity of symptoms among patients and their variability within patients across episodes, two distinct patterns have been discerned in long-term catamnestic studies of schizophrenia patients. First, negative symptoms tend to be less common and severe in the early stages of the illness and to increase in prevalence and severity in the later stages. In the early stages positive symptoms are more likely to dominate the clinical picture. Second, within the constellation of positive symptoms, formed or systematized delusions and hallucinations are more common in the earlier stages of illness, whereas thought disorganization, inappropriate affect, and motor symptoms are more common in the later stages of illness.

Both MRI and MRS offer evidence, which is consistent with a neurodegenerative pathologic process in schizophrenia that occurs primarily but not exclusively in the early stage of the illness. Recent MRI studies of first-episode and childhood-onset schizophrenia samples using more rigorous and standardized methods have found cortical gray matter and ventricular system volume changes. The findings of volume reductions in cortical gray matter and increases in ventricular system volume can be described as consistent with a process causing pathomorphologic progression and neurodegeneration Investigators have considered the role of molecular mechanisms in the neuropathology of schizophrenia. In this context, proponents of neurodegenerative theories have suggested that the absence of gliosis and evidence of cell degeneration could be due to the fact that the pathophysiology involves a graded apoptosis rather than a fulminant necrotic process. Apoptosis is evanescent and difficult to detect histopathologically before or after the process unfolds. Studies have shown that various neurochemical events at the synapse can induce apoptosis. Such triggering actions include excessive glutamate stimulation, calcium influx reactive oxygen species all of that can induce caspase activation in dendrites. Local activation of caspases that initiate the apoptotic cascade can spread to the cell body or remain localized producing neurodegenerative synapse loss and synaptic remodeling. The reduced size and increased density of neurons, in the absence of decreased numbers of neurons or glia and decreased cortical thickness, indicate that cell processes and synaptic connections are reduced in schizophrenia. This is consistent with reports of decreased concentrations of synaptic proteins (e.g., synaptophysin). These cell processes and synapses could be lost as a consequence of a neurochemically mediated (through dopamine and/or glutamate) synaptic apoptosis that would compromise cell function and alter brain morphology without, however, producing serious cell injury (and thus inducing glial reactions).

Although some authors have suggested that pharmacologic treatment suppresses the symptoms of schizophrenia but does not alter the course of the illness or its potential progression, others have suggested that antipsychotic drugs in fact ameliorate the pathophysiologic process that causes psychotic symptoms and leads to clinical deterioration. Moreover, maintenance treatment studies have demonstrated the prophylactic effect of antipsychotic drugs in preventing relapse; treatment, then, may be responsible for mitigating the course of the illness and producing more favorable outcomes.

Three lines of evidence suggest that the novel neurotransmitter Nitric Oxide (NO) play a central role in pathophysiology of schizophrenia. First, schizophrenia-like syndromes can be induced in humans by phencyclidine (PCP), a drug with marked psychomimetic properties. Recent studies indicate that the behavioral and biochemical effects of PCP in rats are blocked by Nitric Oxid synthase (NOS) inhibitors, suggesting that NO plays an important role in the pharmacological effects of PCP. Second, Postmortem brain tissue obtained at autopsy from schizophrenia and control demonstrate increased in NOS in the cerebellum and brainstem of schizophrenic patients. Third, NO play a role in learning and memory, which severly impaired in schizophrenia.

Minocycline is a second-generation tetracycline used in humans, which effectively crosses the blood-brain barrier. Minocycline is commonly used by humans, because of its beneficial ant-imicrobial and anti-inflammatory properties. In addition, it has remarkable neuroprotective qualities in animal models of cerebral ischemia, traumatic brain injury, and Huntington's and Parkinson's disease. The neuroprotective effect of Minocycline is associated with marked inhibition of inducible NO synthase (iNOS), caspase 1 and caspase 3 expression, and p38 mitogen activated protein kinase (MAPK). Recently, it was found that Minocycline also inhibits cytochrome c release and delays progression of amyotrophic lateral sclerosis in mice.

Because Minocycline may inhibit members of the caspase family, the MAP kinase pathway and NOS (which play central role in the neuroprotective effects of Minocycline in different model of brain-disease), we would like to test the neuroprotective effect of Minocycline in the early development (i.e.- at the first psychotic episode) of schizophrenia. The safety record of Minocycline and its ability to penetrate the blood-brain barrier are well known. Therefore, if this drug will be found to have neuroprotective effect in schizophrenia it may be a novel therapy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-35 years;
2. current DSM-IV diagnosis of schizophrenia confirmed by the Structured Clinical Interview for DSM-IV (SCID) conducted by a trained psychiatrist.
3. being at an early phase of the disorder (i.e., within five years of their first exposure to neuroleptic treatment;18)
4. did not receive antipsychotic treatment for six months preceding current symptom exacerbation;
5. baseline total score of more than 60 on the Positive and Negative Syndrome Scale (PANSS).
6. Initiation of treatment with atypical antipsychotic medication equal or less than 14 days prior to study entry (risperidone, olanzapine, quetiapine, or clozapine; 200-600 mg/day chlorpromazine equivalent doses);
7. able to comprehend the procedure and aims of the study.

Exclusion Criteria:

1. acute, unstable, significant or untreated medical illness beside schizophrenia;
2. pregnant or breast-feeding females;
3. A DSM-IV diagnosis of substance abuse or dependency;
4. Known contraindication to minocycline treatment.
5. Treatment with minocycline or Beta-lactam antibiotics in the preceding half year before study entry.
6. Under compulsory hospitalization.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Scale for Assessment of Negative Symptoms (SANS) | Change in SANS scores over the 6-month study

SECONDARY OUTCOMES:
PANSS, CGI, CDS, ITAQ, CANTAB measures, adverse events. | Change during the 6-month duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel - Levkovitz, M.D. PhD., Principal Investigator — Shalvata Mental Health Center
Locations (1):
- The Emotion-Cognition Research Center, The Shalvata Mental Health Care Center, P.O.B. 94., Hod HaSharon, Israel

REFERENCES:
- [Derived] Levkovitz Y, Mendlovich S, Riwkes S, Braw Y, Levkovitch-Verbin H, Gal G, Fennig S, Treves I, Kron S. A double-blind, randomized study of minocycline for the treatment of negative and cognitive symptoms in early-phase schizophrenia. J Clin Psychiatry. 2010 Feb;71(2):138-49. doi: 10.4088/JCP.08m04666yel. Epub 2009 Nov 3. PMID 19895780
- See also: Stanley Research Foundation (SMRI)- grants — http://www.stanleyresearch.org/